CLINICAL TRIAL: NCT05978180
Title: Prospective, Multicenter, Randomized, Parallel Groups Study Comparing the Safety and the Efficacy of the Administration of One Intra-articular Injection of 4.8 ml (HO-1) or Three Intra-articular Injections of 2.2 ml (HS-3) of Pandora Gel to One Intra-articular Injection of 2.5 ml (SINOVIAL®ONE), in Symptomatic Gonarthrosis
Brief Title: Safety of Use and Efficacy of Pandora for Patients Suffering From Gonarthrosis (PANDORA2)
Acronym: PANDORA2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Labrha (Industry)
Collaborators: Statitec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-A00547-38
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Viscosupplementation; Hyaluronic acid; Knee; Intra-articular injection; Tranexamic acid
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, controlled, single blind, randomized in parallel groups Clinical Investigation.
  Subjects will receive one of three viscosupplementations depending on the randomization.
  The study includes two periods :
  * The first period (26 weeks) : prospective, multicenter, randomized in three parallel groups study, comparing the two forms of Pandora gel (HO-1 and HS-3) to SINOVIAL® ONE. The comparison between HO-1 and SINOVIAL® ONE is realized in single blind and the comparison between HS-3 and SINOVIAL® ONE is realized without masking.
  * The second period (26 weeks) is an exploratory, prospective, multicenter phase comparing these same devices without masking.
Who Masked: Participant
Masking Description: Single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Medical Device : HO-1 (Experimental): Single injection Hyaluronic acid associated with tranexamic acid 4.8 ml will be injected in one time Intra-articular single injection
  * Both groups will receive their first injection after a selection visit ; first injection will be planned between 7 days to 30 days after to confirm the enrollment.
  * The injection will be performed at Day 1.
  Interventions: Device: Medical Device : HO-1
- Medical Device : HS-3 (Experimental): Three injections Hyaluronic acid associated with tranexamic acid 2.2 ml will be injected in three times (one injection per week) Intra-articular single injection
  * Both groups will receive their first injection after a selection visit ; first injection will be planned between 7 days to 30 days after to confirm the enrollment.
  * The injections will be performed at Days 1, 8 and 15.
  Interventions: Device: Medical Device : HS-3
- Medical Device : SINOVIAL® ONE (Active Comparator): Hyaluronic acid 2.5 ml will be injected in one time Intra-articular single injection
  * Both groups will receive their first injection after a selection visit ; first injection will be planned between 7 days to 30 days after to confirm the enrollment.
  * The injection will be performed at Day 1.
  Interventions: Device: Medical Device : SINOVIAL® ONE

INTERVENTIONS:
Device: Medical Device : HO-1 — The injection will be performed at Day 1.
  Other Names: Intra-articular single injection
  Arms: Medical Device : HO-1
Device: Medical Device : HS-3 — The three injections will be performed at Days 1, 8 and 15.
  Other Names: Intra-articular three injections
  Arms: Medical Device : HS-3
Device: Medical Device : SINOVIAL® ONE — The injection will be performed at Day 1.
  Other Names: Intra-articular single injection
  Arms: Medical Device : SINOVIAL® ONE

SUMMARY:
The knee osteoarthritis is a frequent degenerative condition that mainly affects subjects over 60, population often weakened by numerous comorbidities and concomitant treatments, justifying the development of new therapies.

The viscosupplementation is a symptomatic treatment for knee osteoarthritis ; the objective of this intra-articular injection of hyaluronic acid is to reduce knee pain and improve mobility. In practice, there are two protocols to administer viscosupplementation : in a single injection or in three injections performed weekly.

The present clinical investigation has the objective to evaluate the safety and efficacy of use of Pandora, a hyaluronic acid associated with tranexamic acid, in a single injection (HO-1) or in three injections performed weekly (HS-3), compared to a referred and commercialized medical device.

DETAILED DESCRIPTION:
This clinical investigation is a prospective, multicenter, randomized, parallel groups study of a class III Medical Device.

This study is designed to compare the safety of use and the efficacy of Pandora in its two forms : in a single injection (HO-1) or in three injections (HS-3) to a single intra-articular injection of 2.5 ml (SINOVIAL®ONE)

A descriptive analysis will be carried out to characterize the demographic data, the history of the disease and its treatments, the clinical and radiological data of the patients at inclusion.

The efficacy of Pandora will be demonstrated by describing the variation of WOMAC A1 score "walking pain" of target knee in repeated measures.

In total, 252 participants will be enrolled across 40 study centers in France and Monaco.

The total duration of subjects' participation is 12 months ; overall study duration including the enrollment period is expected to take approximately 24 months.

ELIGIBILITY:
Inclusion Criteria :

* Patient aged between 35 and 85 years.
* Body mass index (BMI) < 35 kg.m2.
* Medial or lateral femoro-tibial knee osteoarthritis, diagnosed according to the American College of Rheumatology criteria, radiological stage 2 and 3 according to the Kellgren-Lawrence criteria modified by Felson on an X-ray, of the knee in extension, less than 6 months old.
* Knee osteoarthritis responsible for walking pain in the target knee, assessed between 4 and 8 inclusive on an 11 points numerical scale (0 = none to 10 = extreme).
* Unilateral or bilateral knee osteoarthritis if the walking pain in the contralateral knee is < 3 based on 11 points numerical scale (0-10).
* Ambulatory patient able to walk 50 meters without a cane, crutch or walker.
* Patient giving his informed consent.
* Patient agreeing to follow-up study visits.
* Patient affiliated to the health social security system or beneficiary of such plan.
* Patient requiring viscosupplementation according to the investigator.

Exclusion Criteria :

* Patient presenting knee osteoarthritis without impingement joint space narrowing of the femoro-tibial compartment (modified Kellgren stage 0-1) or with complete impingement joint space narrowing on the knee weight-bearing radiograph in extension (modified Kellgren stage 4).
* Patient with bilateral symptomatic gonarthrosis with walking pain of contralateral knee > 3.
* Patient with stage 4 patello-femoral osteoarthritis associated with femoro-tibial osteoarthritis.
* Patient with a flare of osteoarthritis of the target or contralateral knee.
* Patient who received viscosupplementation or Platelet Rich Plasma (PRP) injection, in the target knee, in the 6 months prior to inclusion.
* Patient who received an intra-articular injection of corticosteroids in the target knee in the 2 months prior to inclusion.
* Patients with a skin condition or a wound next to or near the injection site.
* Patients refusing to discontinue treatment with NSAIDs or cox-2 inhibitors during the follow-up period.
* Patient receiving treatment with level III analgesics (strong opioids).
* Patients receiving treatment with diacerhein, avocado and soy unsaponifiables, glucosamine or chondroitin initiated less than 2 months prior to inclusion.
* Patient with hypersensitivity to hyaluronic acid or tranexamic acid.
* Patient with a history of seizures.
* Patient who had arthroscopy of the target knee or major trauma to the target knee during the 3 months preceding inclusion.
* Patient scheduled to undergo surgery, for any cause, of the target knee or other joint of the lower limbs, planned within 6 months of inclusion, likely to interfere with follow-up or evaluation of the patient in the study.
* Patient with Fibromyalgia.
* Patient with an active neurological or vascular musculoskeletal disorder (such as rheumatoid arthritis, lupus, psoriatic arthritis, spondyloarthritis or any other autoimmune disease, Paget's disease, gout, coxopathy, tendinopathy of the lower limb, sciatic or crural radiculalgia) which, in the opinion of the investigator, would be likely to disrupt regular monitoring and/or interfere with the measurement of evaluated knee treatment efficacy.
* Patient with serious hemostasis disorders, venous or lymphatic stenosis of the lower limbs, history of thromboembolic disease - phlebitis or pulmonary embolism - or a high risk of thromboembolism.
* Patients with renal insufficiency.
* Patients with all evolving general condition as cardiac, digestive, endocrine, haematological or broncho-pulmonary which, in the opinion of the investigator, would be likely to disrupt regular monitoring and/or interfere with the measurement of evaluated knee treatment efficacy.
* Breastfeeding patient, pregnant or wishing to be during the 12 months of the study.
* Patients of childbearing age, sexually active without contraception.
* Patients unable to give personal consent.
* Patients participating or having participated in interventional research and whose follow-up ended within 2 months prior to inclusion.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-11-13 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of the two medical devices containing Pandora gel, HO-1 and HS-3, on walking pain in the target knee, compared to the SINOVIAL® ONE. | 6 months
  Variation of the WOMAC A1 score "walking pain" of the target knee in repeated measures (weeks 4,12 and 26), between the first or single injection and the potential injection at week 26.

SECONDARY OUTCOMES:
To evaluate the efficacy of viscosupplementation by HO-1 and HS-3 on walking pain of the target knee between day 1 and week 12. | 3 months
  Variation of the WOMAC A1 score "walking pain" of the target knee between day 1 and week 12 considering the repeated measures at weeks 4 and 12.
To evaluate the efficacy of viscosupplementation by HO-1 and HS-3 on the pain of the target knee at weeks 4, 12 and 26 and week 12 as well as week 52 for patients who didn't require an injection at week 26. | 12 months
  Variation of the pain on target knee, with repeated measures by WOMAC A score, constituted of 5 questions about knee pain, between day 1 and week 12, day 1 and week 26 as well as between day 1 and week 52 for patients who didn't require an injection of HO-1 at week 26.
To evaluate the efficacy of viscosupplementation by HO-1 and HS-3 on the function of target knee at weeks 4, 12, 26 as well as week 52 for patients who didn't require an injection at week 26. | 12 months
  Variation of the function , with repeated measures by the WOMAC C constituted of 17 questions, between day 1 and week 4, day 1 and week 12, day 1 and week 26 as well as between day 1 and week 52 for patients who didn't require an injection at week 26.
To evaluate the efficacy of viscosupplémentation by HO-1 and HS-3 on the analgesic drug consumption at weeks 4, 12, 26 as well as week 52 for patients who didn't require an injection at week 26. | 12 months
  Evaluation by the patient of his analgesic drug consumption during the two weeks prior each visit.
To determine the number (and percentage) of patients "OMERACT-OARSI responsive" at weeks 4,12,26 as well as week 52 for patients who didn't require an injection at week 26. | 12 months
  Number (%) of "responsive" patients according to OMERACT OARSI criterion, at weeks 4, 12 and 26 (and week 52 for patients who didn't require an injection at week 26).
To determine the number (and percentage) of "highly responsive" patients at weeks 4, 12 and 26 as well as week 52 for patients who didn't require an injection at week 26. | 12 months
  Number (%) of "highly responsive" patients with a decrease of WOMAC A1 > 50% at weeks 4, 12 and 26 (and week 52 for patients who didn't have HO-1 injection at S26).
To determine the number (and percentage) of patients in whom target knee pain is considered acceptable according to the PASS criterion at weeks 4,12 and 26 as well as week 52 for patients who didn't require an injection at week 26. | 12 months
  Number (%) of patients reaching the threshold of PASS at weeks 4, 12 and 26 (and week 52 for patients who didn't require an injection at week 26).
To determine the number (and percentage) of patients in whom the decrease of the target knee pain is considered important (MCII criterion) at weeks 4,12 and 26 as well as week 52 for patients who didn't require an injection at week 26. | 12 months
  Number (%) of patients whom the improvement at weeks 4, 12 and 26 (and week 52 for patients who didn't require an injection at week 26), is superior to the MCII.
To determine the number (and percentage) of patients requiring a new injection at S26. | 6 months
  Number (%) of patients requiring an injection of HO-1 at week 26.
To evaluate, at S52, the efficacy of the additional injection of HO-1 at S26 on pain and function of the target knee. | 12 months
  Variation of WOMAC between week 26 and week 52 at patients receiving injection of HO-1 at week 26.
To evaluate, at S52, the benefit of the additional injection of HO-1 at S26 on analgesic drug consumption. | 12 months
  Decrease of analgesic drug consumption between week 26 and week 52 at patients receiving injection of HO-1 at week 26.
To measure the self-reported treatment efficacy by the patient at weeks 4, 12, 26 and 52. | 12 months
  Evaluation of the efficacy of the treatment by the patient based on a 11 points numerical scale (0-10) at weeks 12,26 and 52.
To evaluate the local tolerability (at the target knee), after each injection of HO-1 and HS-3, compared to SINOVIAL® ONE. | 1 month
  Number of adverse events occurring, at the target knee, after each injection during the 4 weeks following the first or only one injection, whose treatments causality is not evaluated as "not related".
To evaluate the global tolerability of HO-1 and HS-3 throughout the follow-up between day 1 and week 52 in comparison with SINOVIAL® ONE. | 12 months
  Number of adverse events occurring during the 52 weeks of follow up, whose treatments causality is not evaluated as "not related".
To assess patient's satisfaction regarding tolerability of HO-1 and HS-3 treatment between day 1 and week 4, compared to SINOVIAL® ONE. | 1 month
  Subjective assessment of tolerability by the patient, based on a 5 points numerical scale, 0 corresponding to "Very Good" and 4 "Very Bad" at day 8, day 15 and week 4 for group's patients HO-1 and SINOVIAL® ONE.
To assess patient's satisfaction regarding the tolerability of HO-1 treatment at week 27 for patients who received an injection at week 26. | 6 months and one week (=27 weeks)
  Subjective assessment of tolerability by the patient, based on a 5 points numerical scale, 0 corresponding to "Very Good" and 4 "Very Bad" at week 27 for patients receiving injection of HO-1 at week 26.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Sac-Epee, Study Director — Labrha; Jean-Charles Balblanc, Dr, Principal Investigator — Hôpital Nord Franche-Comté, HNFC
Locations (35):
- France (34):
  - Cabinet de Rhumatologie, Annecy
  - Centre de Chirurgie Orthopédique du Beaujolais, Arnas
  - Centre de Médecine du Sport du Beaujolais, Arnas
  - Cabinet de Rhumatologie, Bagnols-sur-Cèze
  - Cabinet de Rhumatologie La Savoureuse, Belfort
  - Hôpital Nord Franche Comté, Belfort
  - Cabinet de Rhumatologie de Palente, Besançon
  - Centre de Rhumatologie Nord Isère, Bourgoin
  - Cabinet de Rhumatologie, Castelnaudary
  - Polyclinique des Alpes du Sud, Gap
  - Cabinet de Rhumatologie, Gourdon
  - Centre Médical Dulac, La Ciotat
  - Cabinet Médical Tilsitt, Lyon
  - Centre Orthopédique Santy, Lyon
  - Clinique de la Sauvegarde, Lyon
  - Clinique Saint Charles, Lyon
  - Centre Médico-Social du Lac, Mantes-la-Jolie
  - Cabinet Médical Borely Mermoz, Marseille
  - Cabinet de Rhumatologie, Mâcon
  - Cabinet Médical, Montélimar
  - Groupe Médical Adhémar, Montélimar
  - Cabinet de Rhumatologie, Montpellier
  - Centre Médical Saint Roch, Montpellier
  - Cabinet Médical Pluridisciplinaire Wallach, Mulhouse
  - Cabinet de Rhumatologie, Nîmes
  - Clinique du Ter, Ploemeur
  - Cabinet Médical, Puyricard
  - Cabinet de Rhumatologie, Roanne
  - Cabinet Médical, Saint-Paul-lès-Dax
  - Groupe Médical Spécialisé - Le Premium, Strasbourg
  - Groupe Hospitalier de la Haute Saône - Hôpital de Vesoul, Vesoul
  - Cabinet de Rhumatologie, Villeurbanne
  - Cabinet de Rhumatologie, Viry-Châtillon
  - Pôle de santé des Sept Chemins, Vourles
- IM2S, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sellam J, Courties A, Eymard F, Ferrero S, Latourte A, Ornetti P, Bannwarth B, Baumann L, Berenbaum F, Chevalier X, Ea HK, Fabre MC, Forestier R, Grange L, Lellouche H, Maillet J, Mainard D, Perrot S, Rannou F, Rat AC, Roux CH, Senbel E, Richette P; French Society of Rheumatology. Recommendations of the French Society of Rheumatology on pharmacological treatment of knee osteoarthritis. Joint Bone Spine. 2020 Dec;87(6):548-555. doi: 10.1016/j.jbspin.2020.09.004. Epub 2020 Sep 12. PMID 32931933
- [Background] Balazs EA. Viscosupplementation for treatment of osteoarthritis: from initial discovery to current status and results. Surg Technol Int. 2004;12:278-89. PMID 15455338
- [Background] Concoff A, Sancheti P, Niazi F, Shaw P, Rosen J. The efficacy of multiple versus single hyaluronic acid injections: a systematic review and meta-analysis. BMC Musculoskelet Disord. 2017 Dec 21;18(1):542. doi: 10.1186/s12891-017-1897-2. PMID 29268731
- [Background] Diracoglu D, Tuncay TB, Sahbaz T, Aksoy C. Single versus multiple dose hyaluronic acid: Comparison of the results. J Back Musculoskelet Rehabil. 2016 Nov 21;29(4):881-886. doi: 10.3233/BMR-160714. PMID 27257981
- [Background] Bhadra AK, Altman R, Dasa V, Myrick K, Rosen J, Vad V, Vitanzo P Jr, Bruno M, Kleiner H, Just C. Appropriate Use Criteria for Hyaluronic Acid in the Treatment of Knee Osteoarthritis in the United States. Cartilage. 2017 Jul;8(3):234-254. doi: 10.1177/1947603516662503. Epub 2016 Aug 10. PMID 28618868
- [Background] Li J, Liu R, Rai S, Ze R, Tang X, Hong P. Intra-articular vs. intravenous administration: a meta-analysis of tranexamic acid in primary total knee arthroplasty. J Orthop Surg Res. 2020 Dec 2;15(1):581. doi: 10.1186/s13018-020-02119-1. PMID 33267906
- [Background] Ng W, Jerath A, Wasowicz M. Tranexamic acid: a clinical review. Anaesthesiol Intensive Ther. 2015;47(4):339-50. doi: 10.5603/AIT.a2015.0011. Epub 2015 Mar 23. PMID 25797505
- [Background] Jules-Elysee KM, Tseng A, Sculco TP, Baaklini LR, McLawhorn AS, Pickard AJ, Qin W, Cross JR, Su EP, Fields KG, Mayman DJ. Comparison of Topical and Intravenous Tranexamic Acid for Total Knee Replacement: A Randomized Double-Blinded Controlled Study of Effects on Tranexamic Acid Levels and Thrombogenic and Inflammatory Marker Levels. J Bone Joint Surg Am. 2019 Dec 4;101(23):2120-2128. doi: 10.2106/JBJS.19.00258. PMID 31800425